CLINICAL TRIAL: NCT03056365
Title: Advanced Nurses vs. General Practitioners for the Management of Outpatient Alcohol Detoxification: a Randomized Clinical Trial Comparing Safety and Costs
Brief Title: Advanced Nurses vs. General Practitioners for the Management of Outpatient Alcohol Detox: a Safety and Cost Comparison
Acronym: SAMBA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015_09; 2015-A01936-43 (Other: ID-RCB number, ANSM); PREPS_14-0209 (Other: PREPS number, DGOS)
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2019-02

CONDITIONS: Alcohol Dependence
Keywords: Detoxification; Outpatient; Advanced Nursing; Health Services
MeSH Terms: conditions — Alcoholism | interventions — General Practitioners

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Nurse (AN) (Experimental): The outpatient detoxication procedure will be entirely managed by an advanced nurse team, using a predefined protocol decision algorithm. The protocol allows that the AN team autonomously manages the diazepam dosing during the detox period. Addiction physicians only intervenes in case of severe withdrawal symptoms or serious adverse events.
  Interventions: Procedure: Advanced Nurse (AN)
- General Practitioner (GP) (Active Comparator): The outpatient detoxication procedure is entrusted to a GP who will manage patients and diazepam dosing as he/she thinks best ("as usual" control group)
  Interventions: Procedure: General Practitioner (GP)

INTERVENTIONS:
Procedure: Advanced Nurse (AN) — Protocoled AN-based management of detox
  Arms: Advanced Nurse (AN)
Procedure: General Practitioner (GP) — 'As usual' medical management of detox
  Arms: General Practitioner (GP)

SUMMARY:
The SAMBA study aims to assess the safety and cost comparison of the management of outpatient alcohol detoxification, between an advanced nurse protocol on the one hand (experimental group), and a GP-based treatment on the other hand (standard-of-care group).

In the advanced nurse (AN) group, nurses manage alcohol detox using a predefined protocol based on both the Cushman and CIWA-Ar scales. Depending on the Cushman and CIWA-Ar scores, which are calculated at every consultation, advanced nurse can adjust the diazepam dosing. In case of any serious adverse event or uncontrolled withdrawal complication, an addiction specialist stands in back-up and can be appealed to decide whether the outpatient detox can be continued or whether the patient has to be hospitalized. In the GP group, GPs can manage patients as they wish.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-Tr criteria for alcohol dependence
* Clinical indication for alcohol detoxification
* Social Insurance
* Signed Consent Form for participation

Exclusion Criteria:

* Previous history of seizures
* previous history of delirium tremens
* acute or chronic liver failure
* contraindication for using diazepam
* average daily alcohol use of 300g of ethanol
* SADQ score of 30 or more
* chronic treatment with baclofen or disulfiram
* current DMS-IV-Tr criteria for major depressive episode, or lifelong history of bipolar or psychotic disorder
* any physical, cognitive, or psychiatric disorder that expose the subjects to enhanced risks (at the discretion of the investigator)
* previous participation in the SAMBA study
* social isolation of homelessness (at the discretion of the investigator)
* pregnancy or breastfeeding
* guardianship or curatorship
* previous participation in a biomedical study over the previous month

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Number of patients considered in failure of outpatient alcohol detoxification period | 15 days
  Hospitalization required (any cause) across the 15 days following the detox start

SECONDARY OUTCOMES:
The total costs for each arm by cost-minimization | during the 15 days of the outpatient alcohol detoxification
  All medical costs (visits, medications, hospitalizations, ambulance,..) resulting from the detoxification management
Number of patients reporting at least one recovery in alcohol consumption | during the 15 days of the outpatient alcohol detoxification
  alcohol consumption obtained from A-TLFB data
Number of patients reporting at least one high alcohol intake | during the 15 days of the outpatient alcohol detoxification
  High alcohol intake defined by consumption of more than 5 standard drinks per day
Number of patients with adverse events | during the 15 days of the outpatient alcohol detoxification

CONTACTS AND LOCATIONS:
Overall Officials: Renaud JARDRI, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (26):
- France (26):
  - CH Beziers, Béziers
  - CH Boulogne, Boulogne
  - CHU Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Csapa Anpaa63, Clermont-Ferrand
  - CHU Créteil, Créteil
  - CH Dunkerque, Dunkirk
  - CHU Grenoble, Grenoble
  - CH Lens - CSAPA Le Square, Lens
  - CSAPA CHRU - Le PARI, Lille
  - CH Limoux, Limoux
  - CSAPA Arc-en-Ciel, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Les Apsyades, Nantes
  - Centre LOGOS, Nîmes
  - CH Perpignan, Perpignan
  - Csapa Anpaa66, Perpignan
  - CH Roubaix, Roubaix
  - CSAPA La Trame - ANPAA59, Roubaix
  - CHU Rouen, Rouen
  - CH du Rouvray, Rouvray
  - CH Alpes-Isère, Saint-Egrève
  - CHU Strasbourg, Strasbourg
  - CH Tourcoing, Tourcoing
  - CH Troyes, Troyes

IPD SHARING:
Plan to Share IPD: Undecided